

6th November 2025

Miss Wang Yi School of Health Sciences Universiti Sains Malaysia 16150 Kubang Kerian, Kelantan. Jawatankuasa Etika Penyelidikan Manusia USM (JEPeM)

Human Research Ethics Committee USM (HREC)

Universiti Sains Malaysia Kampus Kesihatan

16150 Kubang Kerian, Kelantan, Malaysia. Tel.: +609 - 767 3000/2354/2362

Fax. : + 609 - 767 2351 Email : jepem@usm.my

Laman Web : www.jepem.kk.usm.my

www.usm.mv

JEPeM Code: USM/JEPeM/KK/25070591

Protocol Title: Enhancing Stability and Jumping Skills Through Combined Static and Dynamic Balance Training in Female Chinese University-Level Gymnastics Beginners.

Dear Miss.,

We wish to inform you that your study protocol has been reviewed and is hereby granted approval for implementation by the Jawatankuasa Etika Penyelidikan Manusia Universiti Sains Malaysia (JEPeM-USM). Your study has been assigned study protocol code USM/JEPeM/KK/25070591, which should be used for all communications to JEPeM-USM in relation to this study. This ethical approval is valid from 6<sup>th</sup> November 2025 until 5<sup>th</sup> November 2026.

Study Site: Gymnastics Teaching and Research Department of Beijing Sport University, China.

The following researchers are also involved in this study:

- 1. Dr. Marilyn Ong Li Yin
- 2. Dr. Rosniwati Ghafar

The following documents have been approved for use in the study.

1. Research Proposal

In addition to the abovementioned documents, the following technical documents were included in the review on which this approval was based:

- 1. Participant Information Sheet and Consent Form (English version)
- 2. Participant Information Sheet and Consent Form (Chinese version)
- 3. Data Collection Sheet

The list of JEPeM-USM members present during the full board meeting reviewing your protocol is attached.

While the study is in progress, we request you to submit to us the following documents:

- 1. Application for renewal of ethical approval 45 days before the expiration date of this approval through submission of **JEPeM-USM FORM 3(B) 2022: Continuing Review Application Form.**
- 2. Any changes in the protocol, especially those that may adversely affect the safety of the participants during the conduct of the trial including changes in personnel, must be submitted or reported using JEPeM-USM FORM 3(A) 2022: Study Protocol Amendment Submission Form.
- 3. Revisions in the informed consent form using the JEPeM-USM FORM 3(A) 2022: Study Protocol Amendment Submission Form.
- 4. Reports of adverse events including from other study sites (national, international) using the JEPeM-USM FORM 3(G) 2022: Adverse Events Report.
- 5. Notice of early termination of the study and reasons for such using **JEPeM-USM FORM 3(E) 2022.**



- 6. Any event which may have ethical significance.
- 7. Any information which is needed by the JEPeM-USM to do ongoing review.
- 8. Notice of time of completion of the study using **JEPeM-USM FORM 3(C) 2022: Final Report Form.**

Please note that forms may be downloaded from the JEPeM-USM website: <a href="https://jepem.kk.usm.my/">https://jepem.kk.usm.my/</a>

JEPeM-USM is in compliance with the Declaration of Helsinki, International Conference on Harmonization (ICH) Guidelines, Good Clinical Practice (GCP) Standards, Council for International Organizations of Medical Sciences (CIOMS) Guidelines, World Health Organization (WHO) Standards and Operational Guidance for Ethics Review of Health-Related Research and Surveying and Evaluating Ethical Review Practices, EC/IRB Standard Operating Procedures (SOPs), and Local Regulations and Standards in Ethical Review.

Thank you.

"MALAYSIA MADANI"

"BERKHIDMAT UNTUK NEGARA"

Sincerely,

ASSOC. PROF. DR. NAZRI MUSTAFFA

Deputy Chairperson Jawatankuasa Etika Penyelidikan (Manusia) JEPeM Universiti Sains Malaysia



Human Research Ethics Committee USM (HREC)

Penyelidikan Manusia USM (JEPeM)

Universiti Sains Malaysia Kampus Kesihatan

Jawatankuasa Etika

16150 Kubang Kerian, Kelantan, Malaysia. Tel.: +609 - 767 3000/2354/2362

Fax. : + 609 - 767 2351 Email : jepem@usm.my

Laman Web: www.jepem.kk.usm.my

www.usm.my

Date of meeting : 2<sup>nd</sup> September 2025 Venue : Through WEBEX Application Time : 9.00 a.m – 2.00 p.m

Meeting No : 716 Panel : Panel C

Members of Committee of the Jawatankuasa Etika Penyelidikan (Manusia), JEPeM Universiti Sains Malaysia who reviewed the protocol/documents are as follows:

| | Member<br>(Title and Name) | Occupation<br>(Designation) | Male/<br>Female<br>(M/F) | Tick (√) present<br>during review<br>process |
|---|---|---|---|---|
| <b>Deputy Chairperson:</b><br>Assoc. Prof. Dr. Nazri Mustaffa | | Deputy Chairperson of Jawatankuasa Etika<br>Penyelidikan (Manusia), JEPeM USM | M | √<br>(Deputy<br>Chairperson) |
| Advisor:<br>Madam Siti Hawa Ali | | Advisor of Jawatankuasa Etika<br>Penyelidikan (Manusia), JEPeM USM | F | √<br>(Advisor) |
| Member Secretary:<br>Dr. Surini Yusoff | | Member Secretary of Jawatankuasa Etika<br>Penyelidikan (Manusia), JEPeM USM | F | √<br>(Member<br>Secretary) |
| Secretary:<br>Mr. Mohd Bazlan Hafidz Mukrim | | Senior Science Officer | М | ✓ |
| Secretariat:<br>Mr. Mohammad Haris Amirul Mohd Yusoff | | Assistant Administrative Officer | M | <b>*</b> |
| Memb | | | | I |
| 1. | Mr. Khairul Ithma Mahdi | Senior Assistant Registrar, Division of<br>Students Development Affairs & Alumni,<br>Health Campus | M | <b>✓</b> |
| 2. | Assoc. Prof. Dr. Md Salzihan Md<br>Salleh | Lecturer, School of Medical Sciences | М | <b>*</b> |
| 3. | Dr. Munirah Mohd Adnan | Lecturer, School of Dental Sciences | F | ✓ |
| 4. | Prof. Dr. Oleksandr Krasilshchikov | Scientific, Non-Institutional Member | M | <b>✓</b> |
| 5. | Dr. Soo Kah Leng | Lecturer, School of Health Sciences | F | ✓ |
| 6. | Dr. Wan Aireene Wan Ahmed | Lecturer, School of Medical Sciences | F | <b>✓</b> |
| 7. | Dr. Wan Mohd Nazlee Wan Zainon | Medical Officer, Hospital Pakar Universiti<br>Sains Malaysia | М | <b>✓</b> |
| 8. | Assoc. Prof. Dr. Norsarwany<br>Mohamad | Lecturer, School of Medical Sciences | F | <b>✓</b> |
| 9. | Dr. Maizura Murad | Lecturer, School of Industrial Technology | F | ✓ |

Jawatankuasa Etika Penyelidikan (Manusia), JEPeM-USM is in compliance with the Declaration of Helsinki, International Conference on Harmonization (ICH) Guidelines, Good Clinical Practice (GCP) Standards, Council for International Organizations of Medical Sciences (CIOMS) Guidelines, World Health Organization (WHO) Standards and Operational Guidance for Ethics Review of Health-Related Research and Surveying and Evaluating Ethical Review Practices, EC/IRB Standard Operating Procedures (SOPs), and Local Regulations and Standards in Ethical Review.

ASSOC. RROF. DR. NAZRI MUSTAFFA

Deputy Champerson Jawatankuasa Etika Penyelidikan (Manusia), JEPeM Universiti Sains Malaysia